CLINICAL TRIAL: NCT05981261
Title: Comparing Pain Intensity and Discomfort in Patients With Parkinson´s Disease and Healthy Controls During Inducement of Mechanical, Thermal, and Chemical Experimental Pain
Brief Title: Experimental Pain in Parkinsons
Acronym: ExPainPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Experimental pain in PD
Record Dates: First submitted 2023-06-09; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-06

CONDITIONS: Pain; Parkinson Disease
MeSH Terms: conditions — Pain; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a within-subject design where each participant is exposed to experimental pain in infraspinatus muscle, gluteus medius muscle, and tibialis anteior muscle in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental pain (Other): Experimental pain
  Interventions: Other: inducement of experimental pain

INTERVENTIONS:
Other: inducement of experimental pain — Inducement of experimental pain

SUMMARY:
Study comparing pain intensity and discomfort in patients with Parkinson´s disease and healthy controls during inducement of mechanical, thermal, and chemical experimental pain

DETAILED DESCRIPTION:
Project: Inducing experimental muscle pain in healthy volunteers, patients with Parkinson's disease in levodopa treatment, and patients with Parkinson's disease with deep brain stimulation treatment

Research team:

* Andrea S. Poulsen (PI), PhD-student, AU
* Sophie Rosenkjær, PhD-student, AU
* Lene Vase, Professor, AU
* Nanna B. Finnerup, Professor, AUH
* Mette Møller, Leading doctor, AUH
* Erisela Qerama Montvilas, Clinical lector, AUH
* Jan Rosner, Post-doc, AUH

Objective: Comparing induced pain levels in (1) healthy volunteers, (2) patients with Parkinson's disease in levodopa treatment, and (3) patients with Parkinson's disease with deep brain stimulation treatment

Participants: 21 healthy volunteers, 21 patients with Parkinson's disease in levodopa treatment, and 21 patients with Parkinson's disease with deep brain stimulation treatment will be recruited from the Department of Neurology at Aarhus University Hospital. Furthermore, recruitment sheets will be posted at Aarhus University Hospital, at Parkinsonforeningen's webpage (https://www.parkinson.dk/) and newsletter and in local newspapers. A power calculation for a Wilcoxcon-Mann-Whitney rank sum test (Three groups) determine 21 in three test groups is adequate (effect size= 0.8; 1-β=.80; α=.05).

Design:Between-subject randomized study where each participant will complete a ≈1 ½ hour test session at the Department of Neurophysiology, Aarhus University Hospital, Denmark. Each test session will include assessment of ongoing pain, experimental pain (thermal, mechanical, and chemical), and motor response latencies.

Procedure: Each test session proceeds as follow: First, participant is greeted in the entry hall at AUH and escorted to the examination room. Investigator goes through test procedures and introduce to assessments. Participant complete measures of ongoing pain followed by assessment of motor response latencies. Then, assessments of thermal heat detection, pain thresholds and pain-autonomic interactions on volar forearm. Next, sites of inducement of mechanical and chemical pain (randomized gluteus medius muscle, tibialis anterior muscle, and infraspinatus muscle) will be identified by use of manual palpation and defined by distinct anatomical landmarks marked with a pen. For each site: assessment of mechanical pain threshold followed by evaluation of intensity and discomfort during pain suprathreshold. Then, inducement of chemical pain by use of hypertonic saline injections. Immediately after injection, evaluation of pain intensity and discomfort followed by assessment of sensory and affective verbal descriptions of pain and patient drawings of pain size and distribution. Finally, measures of pain intensity and discomfort during mechanical suprathreshold pressure on site of injection. There will be a 15 minutes interval between inducement of experimental pain in the three sites for the pain to cease. Investigator escorts participant to the entry hall and thank participant for taking part in the study.

ELIGIBILITY:
Inclusion criteria

* Group healthy volunteers: healthy subjects with no PD diagnosis
* Group PD patients levodopa: Include PD patients treated with levodopa
* Group PD patients DBS: Include PD patients with DBS Exclusion criteria
* Known other neurological or medical disorders (e.g., stroke, neuropathy, diabetes) or other disorders with expected influence on experimental pain
* Known dementia (a score <24 on the MoCA)
* Known untreated depression (a score ≥15 on the Beck Depression Inventory)
* Unable to cooperate
* Treated with painkillers except paracetamol and NSAID (except if pain and treatment is ad-equately stable as evaluated by a doctor)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Thermal induced heat pain | Immediately after assessment of ongoing pain (15 minutes)
  Thermal heat detection and pain thresholds will be measured following the standardized "Quantitative Sensory Testing" protocol
Mechanical induced pain | Immediately after assessment of thermal induced heat pain (15 minutes)
  Mechanical pain thresholds and suprathresholds will be measured by use of a handhold pressor algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe placed on test muscle (gluteus medius muscle, tibialis anterior muscle, and infraspinatus muscle in a randomized order)
Chemical induced pain | Immediately after assessment of mechanical pain (15 minutes)
  Chemical pain will be induced by an injection of hypertonic saline (HS, 5,8% in 1 ml)
Ongoing pain (Clinical pain in daily life) | After assessment of motor response latencies measure (15 minutes)
  Intensity and discomfort of ongoing pain in gluteus medius muscle, tibialis anterior muscle, and infraspinatus muscle will be assessed by use of 11- point Numeric Rating Scale (NRS)
Ongoing pain (Sensory and affective verbal descriptions of pain and patient drawings) | After assessment of motor response latencies measures (15 minutes)
  Sensory and affective verbal descriptions of pain and patient drawings of pain size and distribution will be measured by use of the short-form McGill Pain Questionnaire (SF-MPQ).
Ongoing pain (Pain in PD) | After assessment of motor response latencies measures (15 minutes)
  Pain in PD will be assessed by King´s Parkinson´s disease pain scale (KPPS)

SECONDARY OUTCOMES:
Motor response latencies measure | Prior to assessment of ongoing pain (3 minutes)
  To control for bias due to reaction time in measures which include participant stop buttons, motor response latencies will be assessed by use of a response box

CONTACTS AND LOCATIONS:
Locations (1):
- aarhus university Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No